CLINICAL TRIAL: NCT02274389
Title: Bedaquiline Patient Registry: Prospective Patient Registry of Patients Exposed to Bedaquiline In the United States
Brief Title: A Prospective Patient Registry of Patients Exposed to Bedaquiline
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR104620; RRA-12028 (Other: Janssen Research and Development, LLC); TMC207TBC4001 (Other: Janssen Research and Development, LLC)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Multi-drug Resistant Tuberculosis
Keywords: Pulmonary Multi-drug Resistant Tuberculosis; Bedaquiline; Sirturo; Observational; Prospective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Bedaquiline Patient Registry (BPR)
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — This is an observational study and participants did not receive any intervention in this study. Participants initiating bedaquiline (BDQ) treatment as decided by healthcare provider, will be prospectively observed.

SUMMARY:
The purpose of this study is to describe the medical indication and utilization of expert medical consultation among participants treated with bedaquiline (BDQ), BDQ susceptibility based on minimum inhibitory concentrations (MICs) reported for baseline and subsequent isolates, BDQ drug utilization data to include dose, duration, past treatment history, past medical history, concomitant medications, and health care site of treatment, drug distribution mechanisms used in the administration of BDQ, patient outcomes (clinical and microbiologic) and adverse events among BDQ-treated participants, including deaths.

DETAILED DESCRIPTION:
This is a prospective (observation of a population for a sufficient number of persons over a sufficient number of years to generate incidence or mortality rates subsequent to the selection of the study group) observational (clinical study in which participants may receive diagnostic, therapeutic, or other types of interventions, but the investigator does not assign participants to specific interventions) study of participants treated with BDQ. Participants will be enrolled by their healthcare provider once the healthcare provider decides to treat with BDQ or after BDQ treatment initiation but prior to observation of any participant outcomes. All participants meeting the inclusion criteria and providing informed consent for participation in the study will be enrolled in this study. The registry enrollment period will be open for 36 months with an additional 24 months BDQ treatment-free follow-up for safety assessment for the last participants enrolled during the 36 months enrollment period. Participants' follow-up data will be collected at each visit from the healthcare provider during the course of BDQ and for an additional 24 months after the last BDQ dose or until the participant is lost to follow-up. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of providing informed consent, which must be obtained prior to collection of any patient outcomes and documented laboratory and clinical variables to meet the study objectives
* Participants who have documented enrollment in the bedaquiline patient registry (BPR) prior to the start of BDQ treatments and documented initiation of BDQ treatment after enrollment
* Participants who have documented initiation of BDQ treatment prior to enrollment and have no documented patient outcomes and documented laboratory and clinical variables to meet the objectives of the study

Exclusion Criteria:

* No specific exclusion criteria will be applied in this study other than those scenarios that follow from the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be drawn from the population of all partIcipants treated with bedaquiline (BDQ) in the United States. All participants meeting registry inclusion criteria will be eligible for inclusion in the BDQ patient registry provided they submit the necessary informed consent for participation.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12-24 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Medical Indication for Bedaquiline (BDQ) Treatment and Frequency of use of Expert Medical Consultation With BDQ | Baseline up to 24 months after last BDQ dose
  Indication for a drug refers to the use of that drug for treating a particular disease. Percentage of participants treated using expert medical consultation will be summarized. Percentage of participants with medical indication for BDQ treatment as reported by the healthcare provider and frequency of use of expert medical consultation in multi-drug resistant tuberculosis (MDR-TB) treatment with BDQ will be reported.
Number of Participants With BDQ Susceptibility Based on Minimum Inhibitory Concentration (MIC) | Baseline up to 24 months after last BDQ dose
  The MIC is the lowest concentration of an antimicrobial that will inhibit the visible growth of a microorganism after overnight incubation. Number of participants whose post-enrollment isolates exhibit at least 4-fold increase in BDQ MIC in comparison to baseline MIC, provided that the post-baseline MIC is greater than 0.25 milligram per milliliter (mg/mL) based on phenotypic methods on solid or liquid media.
Maximum Dose of BDQ | Baseline up to Month 12
  Maximum dose of BDQ used will be reported.
Total Duration of BDQ Treatment | Baseline up to Month 12
  Exposure to BDQ will be determined by documentation by the healthcare provider. Duration of BDQ treatment will be calculated from the initiation and discontinuation dates for BDQ. The initiation date for BDQ drug for each participant will be the drug initiation date as reported by the healthcare provider. The discontinuation date will be defined as the date the drug was stopped as reported by the healthcare provider.
Percentage of Participants with Different Drug Distribution Mechanisms Utilized for Drug Administration | Baseline up to Month 12
  Directly observed therapy short-course (DOTS) combines 5 elements: political commitment; microscopy services; drug supplies; surveillance and monitoring systems; and use of highly efficacious regimens with direct observation of treatment. Percentage of participants with drug distribution mechanisms used and DOT use for drug administration will be reported.
Number of Participants With Clinical and Microbiologic Patient Reported Outcomes | Baseline up to 24 months after last BDQ dose
  The following treatment outcomes will be estimated separately for participants with MDR-TB and participants with non MDR cases or MDR status not documented as per World Health Organization (WHO) Treatment of tuberculosis guidelines: cured, treatment completed, treatment failed, died, lost to follow-up, not evaluated, and treatment success.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 24 months after last BDQ dose
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product and does not necessarily have a causal relationship with the treatment. An SAE is any untoward medical occurrence that meets any of the following conditions: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
Comparison of Rate of Observed Outcomes With Nationally Available Reported Rates | Baseline up to Month 36
  Treatment outcome will be evaluated on basis of following parameters; Treatment Completed:without evidence of failure BUT no record that three or more consecutive cultures taken at least 30 days apart are negative after intensive phase; Treatment Failed:Treatment terminated or need for permanent regimen change of at least two anti-tuberculosis drugs because of: Lack of conversion by the end of the intensive phase, or Bacteriological reversion in the continuation phase after conversion to negative, or Evidence of additional acquired resistance to fluoroquinolones or second-line injectable drugs, or Adverse drug reactions; Died:participant who dies for any reason during course of treatment; Lost to Follow-Up:whose treatment was interrupted for 2 consecutive months or more; Not Evaluated:whom no treatment outcome is assigned (this includes cases "transferred out" to another treatment unit and whose treatment outcome is unknown); Treatment Success:The sum of cured and treatment completed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Raleigh, North Carolina, United States